CLINICAL TRIAL: NCT06123676
Title: Introduction to the Clinical Workflow of Y90-PET-CT Post-therapy Scans to Patients Undergoing Y90-microspheres Radioembolisation Therapy
Brief Title: Introduction of Y90-PET-CT Post Radioembolisation Therapy Scans
Acronym: Y90-PET-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ChristieNHS
Record Dates: First submitted 2023-10-31; First posted 2023-11-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arms (Other): Single arm study
  Interventions: Device: Y90-PET-CT scan

INTERVENTIONS:
Device: Y90-PET-CT scan — 40 min extra PET-CT scan - no extra injection of radiotracer. We image the Y90-microspheres administered to these patients during the therapy
  Other Names: Y90-PET-CT protocol post-therapy scan for patients undergoing 90Y-microspheres or 90Y-radioembolization treatment or SIRT at the Christie NHS Hospital

SUMMARY:
Yttrium-90, attached to microspheres, usually referred to as 90Y-microspheres or Y-90 radioembolisation, can be used in some cases to treat patients with liver tumours or liver metastasis. The treatment aim is to infuse the 90Ymicrospheres into the patient's liver. The microspheres get trapped in the lesions of micro-blood vessels while the yttrium-90, a radioactive compound, delivers radiation doses locally at these sites and damages the diseased cells.

Therapy is performed in such a way the 90Y-microspheres are localised in the tumour areas minimising damage to the healthy liver tissue. This treatment requires many steps involving professionals from different medical disciplines.

Patients are scanned in the nuclear Medicine Department on a gamma camera the day after the treatment. This scan is referred as Y-90 bremsstrahlung-SPECT. This posttherapy scan provides a 3-dimensional (3D) image of the distribution of the therapeutic agent in the patient's abdomen so an assessment of how much of the therapeutic agent has gone to the sites of disease can be performed.

In this research project, the investigators would like to evaluate an alternative post-therapy scan to the one routinely performed on the gamma camera. The alternative scan is done on a PET-CT scanner and is referred to as Y90-PET-CT. This type of scan has been reported to provide improved quality images, providing more accurate information on the distribution of the patients therapeutic dose.

For this research project, the investigators will invite a small number of patients undergoing this therapy to be scanned twice after treatment: with the current post-therapy scan on a gamma camera; and with the newly proposed scan method, Y90-PET-CT. Depending on the outcomes of this project, assessed by an expert panel of radiologists and medical physicists, the investigators will determine whether we will introduce this new scanning method into clinical practice in the future.

DETAILED DESCRIPTION:
The study will be conducted on patients with liver cancer and/or liver metastasis, referred to as 90Y-microspheres radiation therapy or Y-90 radioembolisation. There will be 10 patients recruited. No further radioisotope administration will be performed (please refer to section 7 for full eligibility criteria).

Primary Outcome - Introduce and optimise a Y90-PET-CT protocol post-therapy scan for patients undergoing 90Y-radioembolisation treatment. The Y90-PET-CT scan will be used primarily to confirm the radiotracer delivery to the target lesions. A Y90-PET-CT scan is believed to provide improved quality images compared to a Y90-bremsstrahlung-SPECT scan; hence, more accurate information on the success/failure of the therapy is expected to be obtained when using Y90-PET-CT images.

Secondary Outcomes - Introduce in the department post-therapy dosimetry for Y90-microspheres radioembolisation using the optimised 90Y-PET-CT images obtained from the primary objective. This work will be done following published guidelines for post-therapy dosimetry and using pre-existing and bespoke commercial software applications that perform this task.

The investigators expect the images resulting from 90Y-PET-CT will provide better information about the success or not of the infusion of the 90Y-microspheres into the target areas. 90Y-PET-CT will, in turn, provide a better understanding of post-therapy scans in our department, better management of 90Y-radioembolization patients and the development of improved radioembolization treatment-planning models in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver treatment Y90-Microspheres therapy.
* Male or female
* Aged 18-85 years

Exclusion Criteria:

A participant will not be eligible for inclusion in this study if any of the following criteria apply:

* History of, or suffers from, claustrophobia or participant feels unable to lie flat and still on their back for a period of up to 45 minutes in the scanner;

  o Priority will be given to their current clinical care scan Y-90-bremsstrahlung-SPECT
* In the opinion of the clinical team, they are unlikely to comply with the study protocol and restrictions that it imposes (i.e. patient uncomfortable to withstand a double scan on the day); Female participants of childbearing potential must confirm they are not pregnant (a strict requisite before 90Y-therapy anyway).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical comparison of current post-therapy scans, Y-90-bremsstrahlung-SPECT, with 90Y-PET-CT for a cohort of 10 patients assessing the feasibility of performing only 90Y-PET-CT post-therapy in the future. | 12 months
  The success criterion of this project will be whether the investigators can incorporate 90Y-PET-CT scans in the department in the future. This will be done by directly comparing 90Y-PET-CT scans with Y-90-bremsstrahlung-SPECT images for each patient and also considering the impact of introducing additional PET-CT scans into the clinical workflow in a very busy Nuclear Medicine department.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS - Nuclear Medicine Department, Manchester, United Kingdom